CLINICAL TRIAL: NCT04095533
Title: ICU Associated Weakness and Its Association With Tibialis Anterior Cross-sectional Area Changes Assessed by Serial Bedside Ultrasound Assessments
Brief Title: ICU Associated Weakness and Bedside Ultrasound Assessment
Status: Terminated | Type: Observational
Why Stopped: Coronavirus pandemic halted in-unit enrolment and participation
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB18-1859
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2019-09

CONDITIONS: Sarcopenia; ICU Acquired Weakness
Keywords: critical care
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis: Starting at admission to ICU, patients admitted to a mixed medical-surgical ICU will be assessed every second day to determine their muscle size as measured by ultrasound, and their muscle strength as measured clinically using the Medical Research Council strength assessment at the bedside.
  One-time Measures:
  * Illness severity as measured by the SOFA score within the first 24 hours of admission.
  * duration of mechanical ventilation
  * duration of stay in the ICU
  * duration of stay in the hospital
  Interventions: Other: Tibialis anterior muscle cross-sectional area assessment by ultrasound; Other: Muscle strength assessment

INTERVENTIONS:
Other: Tibialis anterior muscle cross-sectional area assessment by ultrasound — Assessed using bedside ultrasound with repeat assessments every second day up to 2 weeks of ICU admission, or until discharge from ICU to yield an overall rate of muscle area decline reported as a %/day average muscle atrophy rate.
  Tibialis anterior cross-sectional area assessments will be assessed by measurement ultrasound to both legs with portable bedside ultrasound. The cross sectional area will be measured in cm^2 at 5 cm distal to the lateral eminence of the tibial tuberosity along the muscle belly. Image processing will be performed at the bedside using features available on the ultrasound device. Muscle boundaries will be marked on the device and the cross-sectional area (computed from the perimetral contour of the muscle section) will be determined. This process will be repeated for two times for each leg.
Other: Muscle strength assessment — Assessed using clinical bedside evaluation every second day with the Medical Research Council Sum Score. This is a clinical assessment of strength of 6 different muscle groups (shoulder abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and ankle dorsiflexors) on each side of the body and recorded as a score between 0 (flaccid) and 5 (full strength).

SUMMARY:
ICU-associated weakness is a common experience for people following a critical illness. It is associated with important patient and system-relevant outcomes. Diagnosing ICU-associated weakness can be challenging because making the diagnosis relies on volitional participation in strength testing by the patient in a very ill population that is often sedated or restrained.

This study proposes to test if bedside ultrasound of tibialis anterior (a non-invasive test that doesn't require active participation by the patient) correlates with clinical whole-body weakness in critically ill patients admitted to an ICU with sepsis.

DETAILED DESCRIPTION:
BACKGROUND

Physical weakness is a common during and after critical illness. Weakness can develop for multiple reasons, but it can be generally be grouped into three overlapping categories:

1. Nervous system dysfunction - weakness can result from impairments in the nervous system control of muscles;
2. Muscle size reductions (i.e. sarcopenia) - muscles become smaller with disuse, and;
3. Muscle force reductions (i.e. dynapenia) - muscles develop contractile impairments.

In critical care, diagnostic criteria have been developed for a syndrome of weakness called intensive care unit-acquired weakness (ICU-AW). ICU-AW has important clinical implications. It is associated with delayed ventilator weaning, increased mortality, and longer lengths of stay in the hospital. ICU-AW can also have consequences for patients after they leave the hospital. ICU-AW can be implicated in impairments in quality of life and physical function such as difficulty climbing stairs, and delays in returning to work.

Diagnosing ICU-AW is not trivial and it is centered on assessments targeted primarily to assessing dynapenia. The diagnostic criteria are clear but making the diagnosis relies on the active participation of patients, and the reliable subjective assessment by clinicians at the bedside. Factors such as sedation, restraint use, paralytic medications, pain, and dressings can all confound the assessment of a patient's strength.

To augment patient assessments, it is possible that assessments of sarcopenia might be helpful in highlighting who might be at risk for muscle dysfunction in the ICU.

RESEARCH QUESTION AND OBJECTIVES Do serial measurements of tibialis anterior muscle cross-sectional area (a muscle in the leg) using bedside ultrasound correlate with clinical weakness in people admitted to the ICU for sepsis?

Primary Outcome:

Determine if the rates of decline of tibialis anterior muscle cross-sectional areas (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate with bedside clinical measures of strength using the medical research council (MRC) sum score (a score between 0 and 60).

Secondary Outcomes:

Determine if rates of decline of tibialis anterior muscle cross-sectional areas correlate with:

1. Ankle dorsiflexion strength, measured using the Medical Research Council (MRC) Scale for muscle strength (a score between 0 and 5);
2. Illness severity at admission to the ICU, measured by the Sequential Organ Failure Assessment (SOFA) score (a score between 0 and 24);
3. Duration of mechanical ventilation (days),
4. Duration of ICU length of stay (days), and;
5. Duration of hospital length of stay (days).

METHOD Each day, new admissions to a mixed medical-surgical ICU will be screened. Any person admitted with a diagnosis of sepsis will be considered for invitation to the study. Potential participants will be excluded if they are children (age < 18 years), if they have preexisting diagnoses that would plausibly affect the size of the muscles in their leg, or if they have medical conditions that would preclude an assessment of their strength. Participants who are appropriate for inclusion in the study will be approached for informed consent.

For participants who consent, every second day the cross-sectional area of the tibialis anterior muscle bulk on each leg will be measured (cm^2) using bedside ultrasound. These measurements will be accompanied by a clinical assessment of strength using the Medical Research Council (MRC) strength scale on six muscle groups bilaterally (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion). Participants will continue to be evaluated every other day until they leave the ICU, or until their 14th day of admission to the ICU. Chart reviews will supplement these data to allow for the determination of the secondary objectives (e.g. SOFA scores, hospital lengths of stay).

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (age > 18 years);
2. admitted to the ICU with a diagnosis of sepsis, and;
3. an ICU duration of stay of greater than 4 days (two allow for serial assessments of muscle strength and size).

Exclusion Criteria:

1. Any pre-existing diagnosis that would reasonably impact a participant's muscle bulk, strength, coordination, or ability to participate in the assessment

   * Critical illness myopathy, critical illness neuropathy, and critical illness polyneuropathy diagnosed in the current ICU stay are not to be considered exclusion criteria as these diagnoses are directly related to the research question
   * Delirium is not considered an exclusion criteria for this study so long as at least two strength assessments can be performed during the course of the participant's ICU stay.
2. Any activity orders or movement restrictions (including medical devices such as casts or external fixation devices) that would preclude accurate motor strength assessment.
3. Dressings, casts, or medical implements that would preclude or impede ultrasound assessment of tibialis anterior muscle cross-sectional area in both legs.
4. Patients who are "proned" or in positions that make assessing tibialis anterior with ultrasound or physical exam impractical.
5. Re-admission to ICU within the same hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include any adult participants that are admitted to a mixed medical-surgical ICU with a diagnosis of sepsis. There are no restrictions based on the source of the infection (e.g. upper respiratory tract infections vs. abdominal sepsis from a perforated viscous) and no restriction based on the treatment provided (e.g. surgery for source control vs. systemic antibiotics).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Correlation of tibialis anterior muscle atrophy development with whole-body strength | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate with bedside clinical measures of strength using the MRC sum score.

SECONDARY OUTCOMES:
Correlation of tibialis anterior muscle atrophy development with ankle dorsiflexion strength | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate with bedside clinical measures of ankle dorsiflexion strength.
Correlation of tibialis anterior muscle atrophy development with illness severity at admission ICU | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate Illness severity at admission to the ICU, measured by the Sequential Organ Failure Assessment (SOFA) score.
Correlation of tibialis anterior muscle atrophy development with duration of mechanical ventilation in ICU | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate the duration of mechanical ventilation in ICU (days).
Correlation of tibialis anterior muscle atrophy development with ICU length of stay | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate the duration of ICU admission (days).
Correlation of tibialis anterior muscle atrophy development with hospital length of stay | First two weeks of ICU admission
  Determine if the rates of decline of tibialis anterior muscle cross-sectional area (%/day) measured by bedside ultrasound on participants admitted to an ICU for sepsis correlate the duration of hospital admission (days).

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No